CLINICAL TRIAL: NCT06034028
Title: J-Valve TF Early Feasibility Study
Acronym: JVTF EFS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JC Medical, Inc., an affiliate of Edwards Lifesciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JCM-001
Record Dates: First submitted 2023-08-28; First posted 2023-09-13 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Aortic Valve Disease; Aortic Valve Insufficiency; Aortic Regurgitation
Keywords: J-Valve TF System; Transcatheter Aortic Valve Replacement; Transcatheter Aortic Valve Implantation; Transcatheter Heart Valve; Transfemoral; TAVR; TAVI; THV; VHD; Valvular Heart Disease; Valve Disease
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Insufficiency; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- J-Valve TF System (Experimental)
  Interventions: Device: J-Valve TF System

INTERVENTIONS:
Device: J-Valve TF System — The J-Valve TF System is a transcatheter aortic valve replacement system that consists of the J-Valve TF Bioprosthesis, J-Valve TF Delivery Device, and Loading Accessories.

SUMMARY:
The main objective of this study is to assess the preliminary safety and effectiveness of the J-Valve TF System in patients with symptomatic severe native aortic regurgitation who are judged by a multi-disciplinary heart team to be eligible for the device and to be at high risk for open surgical aortic valve replacement.

DETAILED DESCRIPTION:
The EFS is a prospective, single arm, multi-center, interventional study that will enroll up to 25 subjects in up to 15 centers in the United States and/or Canada and report the primary endpoint of all-cause death or disabling stroke at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient has symptomatic (NYHA FC ≥ IIs) severe (≥3+) native AR (per 2020 ACC/AHA Guideline for Management of Patients with Valvular Heart Disease) diagnosed by echocardiography. Patients will be assessed according to the current American Society of Echocardiography Guidelines for Non-invasive Evaluation of Native Valve Regurgitation. Transesophageal echocardiography (TEE) or cardiac MRI (CMR) will be used in case of indeterminant AR;
* Patient is judged by a multi-disciplinary heart team to be at high risk for surgery, based on the ACC/AHA guidelines for management of patients with valvular heart disease: STS-PROM score ≥8%, or if <8%, significant co-morbidities that are not captured by the STS-PROM score (e.g., ≥2 frailty indices, 1 to 2 major organ system compromise, the presence of certain procedure-specific factors that affect surgical mortality), based on the consensus of a multi-disciplinary heart team;
* Patient has suitable anatomy for J-Valve implantation (see anatomic exclusions below);
* Patient or the patient's legal representative has provided written informed consent;
* Patient or patient's legal representative agrees to comply with all required post-procedure follow-up visits.

Exclusion Criteria:

* Patients that are at prohibitive surgical risk (predicted risk for mortality or major morbidity at 30 days >50% with SAVR);
* Mixed aortic valve disease, defined as coexistence of > moderate aortic valve stenosis with severe AR;
* Known hypersensitivity or contraindication to aspirin, heparin, bivalirudin, ticlopidine, clopidogrel, Nitinol (Nickel, Titanium, Aluminum) or sensitivity to contrast media, which cannot be adequately premedicated;
* Blood dyscrasias as defined: leukopenia (WBC <1000 mm3), thrombocytopenia (platelet count <50,000 cells/mm3), history of bleeding diathesis or coagulopathy;
* Active infection, including infective endocarditis;
* Liver failure (Child-C);
* Reduced left ventricular function with left ventricular ejection fraction (LVEF) <25% as measured by resting echocardiogram;
* Uncontrolled atrial fibrillation (e.g., resting heart rate >120 bpm);
* Pregnancy or intent to become pregnant prior to completion of all protocol follow-up requirements;
* Renal insufficiency (eGFR <25) and/or end stage renal disease requiring chronic dialysis;
* Pulmonary Hypertension (systolic pressure ≥2/3 of systemic);
* Severe Chronic Obstructive Pulmonary Disease (COPD) = requiring steroids or requiring continuous home O2
* Severe mitral or severe tricuspid regurgitation or stenosis;
* Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within six weeks of treatment;
* Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support;
* Recent (within 6 months of treatment) cerebrovascular accident (CVA) or transient ischemic attack (TIA);
* Active gastrointestinal (GI) bleeding that would preclude anticoagulation;
* Untreated multivessel coronary artery disease with a Syntax score >22 and/or unprotected left main coronary artery;
* Evidence of acute myocardial infarction within 1 month of intended procedure;
* PCI within 30 days of intended procedure;
* Estimated life expectancy of less than 24 months due to associated (excluding cardiac) co-morbid conditions;
* Left Ventricular Assist Device (LVAD) dependent;
* Participating in another study that may influence the outcome of this study;
* Need for emergency surgery for any reason;
* Previous aortic bioprosthesis or mechanical implant.

Anatomic Exclusion Criteria:

* Ascending Aortic diameter >5 cm;
* Aortic Annulus Perimeter <57 mm or >104 mm;
* Access vessel minimum diameter <5.5 mm;
* LVEDD >75 mm;
* Bicuspid aortic valve disease;
* Congenital univentricle or other condition that, in the opinion of the investigator and/or consulting physician, may constitute an unwarranted surgical risk.
* Abdominal aortic aneurysm ≥ 4.0 cm;
* Aorto-iliac disease requiring intervention to facilitate delivery of access sheath;
* Excessive tortuosity of delivery system pathway, defined as severe tortuosity of multiple vessels including iliofemoral, descending aorta, ascending aorta, aortic arch, and aortic angle >80⁰. In most cases, this exclusion will be identified and assigned following review by the multi-disciplinary Screening Committee.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2029-08-25 (Estimated)

PRIMARY OUTCOMES:
Number of patients that do not experience death or disabling stroke | 30 days after the valve procedure
  Freedom from death or disabling stroke Disabling stroke is evaluated using a standardized scale

SECONDARY OUTCOMES:
Number of patients and procedures achieving technical success | At point patient exits the procedure room
  Procedures achieving the following:
  * Patient is alive;
  * There was successful access, delivery of the valve, and retrieval of the delivery device;
  * There was correct positioning of a single prosthetic heart valve into the proper anatomical location;
  * There was no need for surgery or intervention due to the device, except permanent pacemaker placement, or for a major complication that it vascular, access-related, or cardiac in nature
Number of patients and procedures achieving device success | 30 days after the valve procedure
  * There was successful access, delivery of the valve, and retrieval of the delivery device;
  * There was correct positioning of a single prosthetic heart valve into the proper anatomical location;
  * There was no need for surgery or intervention due to the device, except permanent pacemaker placement, or for a major complication that it vascular, access-related, or cardiac in nature;
  * Patient is alive;
  * There was not surgery or intervention due to the device, except permanent pacemaker placement, or for a major complication that it vascular, access-related, or cardiac in nature;
  * The valve was performing as intended, measured by echocardiography
Number of patients with a safety-related event outcome | 30 days after the valve procedure
  Freedom from:
  * All-cause death;
  * All stroke;
  * Valve Academic Research Consortium (VARC)-3 type 2-4 bleeding;
  * Major vascular, access-related, or cardiac structural complication;
  * Acute kidney injury stage 3 or 4;
  * Moderate or severe aortic regurgitation;
  * New permanent pacemaker due to procedure related conduction abnormalities;
  * Surgery or intervention related to the device.
Number of patients experiencing success | 1 year after the valve procedure
  No re-hospitalization or re-interventions for the underlying condition and improvement, from baseline, in symptoms, which are measured using the Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary (OS) score.
  Success in an increase from baseline of 10 or more points on the KCCQ-OS score.
Number of patients meeting clinical efficacy outcome at 2 years | 2 years after the valve procedure
  * Freedom-from all-cause death;
  * Freedom from all stroke;
  * Freedom from hospitalization for procedure- or valve-related causes;
  * Freedom from KCCQ-OS score < 45 or decline from baseline of >10 points;
  * Good Outcome: Alive with change in KCCQ-OS score >=10 points;
  * Excellent outcome: Alive with change in KCCQ-OS score >=20 points.
Number of patients meeting clinical efficacy outcome at 3 years | 3 years after the valve procedure
  * Freedom-from all-cause death;
  * Freedom from all stroke;
  * Freedom from hospitalization for procedure- or valve-related causes;
  * Freedom from KCCQ-OS score < 45 or decline from baseline of >10 points;
  * Good Outcome: Alive with change in KCCQ-OS score >=10 points;
  * Excellent outcome: Alive with change in KCCQ-OS score >=20 points.
Number of patients meeting clinical efficacy outcome at 4 years | 4 years after the valve procedure
  * Freedom-from all-cause death;
  * Freedom from all stroke;
  * Freedom from hospitalization for procedure- or valve-related causes;
  * Freedom from KCCQ-OS score < 45 or decline from baseline of >10 points;
  * Good Outcome: Alive with change in KCCQ-OS score >=10 points;
  * Excellent outcome: Alive with change in KCCQ-OS score >=20 points.
Number of patients meeting clinical efficacy outcome at 5 years | 5 years after the valve procedure
  * Freedom-from all-cause death;
  * Freedom from all stroke;
  * Freedom from hospitalization for procedure- or valve-related causes;
  * Freedom from KCCQ-OS score < 45 or decline from baseline of >10 points;
  * Good Outcome: Alive with change in KCCQ-OS score >=10 points;
  * Excellent outcome: Alive with change in KCCQ-OS score >=20 points.
Number of patients achieving long-term clinical efficacy for valve function | 5 years after the valve procedure
  Freedom from:
  * Bioprosthetic valve failure (defined as Valve-related mortality or aortic valve re-operation/re-intervention or Stage 3 hemodynamic valve deterioration);
  * Stroke or peripheral embolism (presumably valve- related, after ruling out other non-valve etiologies);
  * VARC-3 Type 2-4 bleeding secondary to or exacerbated by antiplatelet
  * or anticoagulant agents, used specifically for valve- related concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Dean J Kereiakes, MD, Principal Investigator — The Christ Hospital; Michael J Reardon, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (9):
- United States (9):
  - HonorHealth, Scottsdale, Arizona
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Cardiovascular Institute of the South, Houma, Louisiana
  - University at Buffalo, Buffalo, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Houston Methodist Hospital, Houston, Texas
  - Swedish Medical Center Cherry Hill, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Writing Committee Members; Otto CM, Nishimura RA, Bonow RO, Carabello BA, Erwin JP 3rd, Gentile F, Jneid H, Krieger EV, Mack M, McLeod C, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A, Toly C. 2020 ACC/AHA Guideline for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2021 Feb 2;77(4):e25-e197. doi: 10.1016/j.jacc.2020.11.018. Epub 2020 Dec 17. No abstract available. PMID 33342586
- See also: JC Medical, Inc. company website. — http://j-valve.com